CLINICAL TRIAL: NCT03418805
Title: A Randomized, 4-way Crossover Study to Evaluate the Food Effect and the Absorption Profile of Investigational Product of "Ibuprofen Controlled-Release Tablets 600 mg" in Comparison to the Reference Standard Ibuprofen Tablets 200 mg in Normal Healthy Volunteers
Brief Title: To Evaluate the Food Effect and the Absorption Profile of Ibuprofen Controlled-Release Tablets 600 mg in Comparison to the Reference Standard Ibuprofen Tablets in Normal Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's consideration of product development strategies
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OVEIBUZ20151221
Record Dates: First submitted 2018-01-08; First posted 2018-02-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Pain Control
Keywords: Ibuprofen; Controlled-Release; pain control; Healthy Volunteers; Food Effect
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ibuprofen CR Tablet 600 mg-fasting (Experimental): One tablet of IBUCR 600 mg under fasting condition
  Interventions: Drug: Ibuprofen CR Tablets 600 mg
- Ibuprofen CR Tablet 600 mg-fed (Experimental): One tablet of IBUCR 600 mg under fed condition
  Interventions: Drug: Ibuprofen CR Tablets 600 mg
- Advil Ibuprofen table 200 mg-fasting (Active Comparator): IBUAdv with a 4-hour dosing interval for 3 tablets (3×200 mg, q4h) under fasting condition
  Interventions: Drug: Advil Ibuprofen table 200 mg
- Motrin IB Ibuprofen Tablets 200 mg-fasting (Active Comparator): IBUMot with a 4-hour doing interval for 3 tablets (3×200 mg, q4h) under fasting condition
  Interventions: Drug: Motrin IB Ibuprofen Tablets 200 mg

INTERVENTIONS:
Drug: Advil Ibuprofen table 200 mg — Administration of the comparator drug:
  Three tablets (dosing at a 4-hour interval, q4h) of reference ibuprofen standard products, followed by 24 hours after the first dose administration.
  Other Names: Advil® Ibuprofen Immediate-Release Tablet 200 mg
  Arms: Advil Ibuprofen table 200 mg-fasting
Drug: Motrin IB Ibuprofen Tablets 200 mg — Administration of the comparator drug:
  Three tablets (dosing at a 4-hour interval, q4h) of reference ibuprofen standard products, followed by 24 hours after the first dose administration.
  Other Names: Motrin® IB Ibuprofen Tablets 200 mg
  Arms: Motrin IB Ibuprofen Tablets 200 mg-fasting
Drug: Ibuprofen CR Tablets 600 mg — Administration of the investigational product:
  Single oral dose of IBUCR, followed by 28 and 32 hours after the dose administration for fasted and fed studies, respectively
  Other Names: Ibuprofen Controlled-Release Tablet 600 mg
  Arms: Ibuprofen CR Tablet 600 mg-fasting; Ibuprofen CR Tablet 600 mg-fed

SUMMARY:
To evaluate the food effect of Ibuprofen CR Tablets 600 mg (IBUCR), and its bioavailability comparison versus 3 doses of the reference arms including Advil® Ibuprofen Tablets 200 mg (IBUAdv) and Motrin® IB Ibuprofen Tablets 200 mg (IBUMot) in normal healthy volunteers.

DETAILED DESCRIPTION:
This randomized, open label, four-way crossover phase I study is to evaluate the food effect of Ibuprofen CR Tablets 600 mg (IBUCR), and its bioavailability comparison versus 3 doses of the reference arms including Advil® Ibuprofen Tablets 200 mg (IBUAdv) and Motrin® IB Ibuprofen Tablets 200 mg (IBUMot) in normal healthy volunteers.

This study will enroll at least 26 evaluable subjects. The duration for test and reference treatments is 24 to 32 hours with a washout period of at least 5 days after the last dose administration of study drugs. The total study will take at least 28 days.

Subjects who meet all eligible requirements for participating in the study will receive all following interventions according to one of the 4 random sequences by Williams design.

1. One tablet of IBUCR 600 mg under fasting condition
2. One tablet of IBUCR 600 mg under fed condition
3. IBUAdv with a 4-hour dosing interval for 3 tablets (3×200 mg, q4h) under fasting condition
4. IBUMot with a 4-hour doing interval for 3 tablets (3×200 mg, q4h) under fasting condition

The blood sampling schedule are described as follows:

-For subjects receiving IBUCR (fed and fasted): Before dose administration (blank) and at 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 18h, 24h, 28h, 32h post-dose (A total of 17 samples per subject)

-For subjects receiving IBUAdv/IBUMot (fasted): Before dose administration (blank) and at 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 4.5h, 5h, 5.5h, 6h, 6.5h, 7h, 8h, 8.5h, 9h, 9.5h, 10h, 10.5h, 11h, 12h, 16h, 20h, 24h post-dose (A total of 25 samples per subject)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are 20 years of age or older.
2. Subjects whose body mass index (BMI) at screening is within a range of ≧18.5 kg/m2 and <25.0 kg/m2.

   BMI = Body Weight (kg) / [Height (m)]2 And body weight is not less than 50 kg and 45 kg for males and females, respectively.
3. Subject's medical history shows no contraindication to the test medications (hypersensitivity to ibuprofen or any component of test and reference products).
4. Subjects who are judged to be in good health by the investigator based upon the results of physical examinations (PEs), chest X-ray (within 180 days prior to the first dose of the study) and routine laboratory tests.
5. The female subject shows negative pregnancy test results within 30 days prior to the first dose of the study.
6. The Subject did not take any of the following medications in the specified durations:

   * Any medication within 14 days prior to the first dose of the study
   * Any enzyme inducer or inhibitor within 30 days prior to the first dose of the study
7. Subject understood and has signed the written informed consent form.

Exclusion Criteria:

1. Subjects with any properly diagnosed disease within 30 days prior to the first dose of the study.
2. Subjects with a clinically significant hematological, endocrine, cardiovascular, hepatic, renal, gastrointestinal, and/or pulmonary disorder; subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism and excretion of drugs; subjects who has had any previous gastrointestinal surgery, except appendectomy if performed >90 days prior to the first dose of the study
3. Subjects who require treatment with any medications, either prescription or non-prescription (excluding vitamins and food supplements), within 30 days prior to the first dose of the study
4. Subjects who have received any known hepatic or renal clearance-altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazine, clarithromycin, trolearndomycin, ketoconazole, miconazole, fluconazole, itraconazole) for a period of up to 30 days prior to the first dose of the study
5. The subject had participated in investigational drug trials and took any investigational drug within 60 days prior to the first dose of the study.
6. The subject had blood donation more than 250 and 500 mL within 60 and 90 days, respectively prior to the first dose of the study.
7. The subject had a history of drug abuse or alcohol abuse.
8. Subjects cannot stop smoking and caffeine-intakes for 48 hours prior to the first dose of the study and during the entire study period.
9. Subjects who are pregnant or lactating
10. For enrollment of female subjects with child-bearing potential, the subject must be practicing sexual abstinence or be using and willing to continue to use a medically acceptable form of birth control for at least 30 days prior to screening (that period will extend to 3 months for oral contraceptive use) and for at least 30 days after the last dose of study drug. For a subject to be considered not to be of child-bearing potential, she must have been amenorrheic for at least 2 years, or must have had a hysterectomy, a bilateral tubal ligation, and/or a bilateral oophorectomy (as determined by the medical history). The male partner of a female study subject with childbearing potential must use a condom and ensure that his partner uses a suitable method of contraception as outlined above.
11. Subjects who are inappropriate to participate in this study, as judged by the medical investigator or sub-investigator
12. Subjects with any contraindication to the use of test medications
13. Subjects who are carriers of hepatitis B virus, hepatitis C virus, or are syphilis (STS) positive, or human immunodeficiency virus (HIV) positive

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma concentration of the period (AUC0-last) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration at each treatment period (Cmax,tp) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration of the first dosing (Cmax) | 1 month
  Individual ibuprofen plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | 1 month
  Individual ibuprofen plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | 1 month
  Individual ibuprofen plasma concentration-time profile for each treatment period will be established.
Mean residence time (MRT) | 1 month
  Individual ibuprofen plasma concentration-time profile for each treatment period will be established.
The maximum ibuprofen plasma concentration within 1 hour after the first dose administration (Cmax0-1h) | 0.5h and 1h post-dose
  The Cmax0-1h will be observed. The mean Cmax0-1h of test and reference treatments under fasting condition will be calculated. Percentage of the test drug-treated subjects with higher or equal Cmax0-1h compared to that of receiving the reference treatments under fasting condition will be calculated.
The minimum ibuprofen plasma concentration within a time window of 1-12 hours after the first dose administration (Cmin1-12h) | 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 7h, 8h and 12h post-dose
  The Cmin1-12h will be observed. The mean Cmin1-12h of test and reference treatments under fasting condition will be calculated.
The mean time to drop to the Cmin1-12h of reference treatments | 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 18h, 24h, 28h, 32h post-dose
  For the plasma ibuprofen concentration of test treatments under fasting condition, the mean time to drop to the Cmin1-12h of reference treatments will be calculated.
Plasma ibuprofen concentrations at 8-hour (C8h) after the first dose administration | 8-hour after the first dose administration
  The C8h after the first dose administration will be observed (prior to the 8-hour dose administration for the reference treatments). The mean C8h of test and reference treatments under fasting condition will be calculated.
Plasma ibuprofen concentrations at 12-hour (C12h) after the first dose administration | 12-hour after the first dose administration
  The C12h after the first dose administration will be observed. The mean C12h of test and reference treatments under fasting condition will be calculated.
Percentage of the test drug-treated subjects with higher or equal C8h compared to that of receiving the reference treatments (before dose 3) under fasting condition | 1 month
Percentage of the test drug-treated subjects with higher or equal C12h compared to that of receiving the reference treatments under fasting condition | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No